CLINICAL TRIAL: NCT05151354
Title: Attachment as a Moderator of the Relationship Between Patient Self-disclosure and Psychotherapy Outcome: Separating Within- From Between-patient Effects
Brief Title: Attachment, Patient Self-disclosure and Psychotherapy Outcome
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Simone Jennissen, Principal Investigator, University Hospital Heidelberg
Other Study IDs: Attach-Sel-2021
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Psychotherapy; Attachment; Self Disclosure; Treatment Outcome
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychotherapy — Patients receive 8 weeks of inpatient psychotherapeutic treatment. Treatment consists of individual and group psychodynamic psychotherapy, as well as an individual combination of art, music, body-oriented and relaxation therapies, which are also carried out in group settings. Treatments is provided by an interdisciplinary team of psychotherapists with a medical or psychology degree, art of music therapists, social workers, physiotherapists and specialist nurses.

SUMMARY:
This study investigates whether within- and between-patient effects of attachment moderate the association between self-disclosure and psychotherapy outcome.

DETAILED DESCRIPTION:
Participants are recruited at the University Clinic Heidelberg at the beginning of their (usually) 8-week inpatient treatment. After informed consent, patients routinely fill out weekly questionnaires on attachment, self-disclosure, and symptom severity.

This study is the first to disentangle stable, trait-like (between-person) effects of both attachment and self-disclosure from within-person changes over the course of treatment. The study investigates whether (changes in) attachment moderate the association between (changes in) self-disclosure and psychotherapy outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients of at least 18 years of age
* treated at the inpatient unit of a hospital for psychosomatic medicine
* provided measurements of symptoms, attachment style, and self-disclosure for at least one measurement occasion

Exclusion Criteria:

* bipolar, acute psychotic or substance abuse disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients undergoing inpatient treatment at the university hospital Heidelberg.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Symptom Checklist Short Form (SCL-K11) | for each participant: weekly assessment for 8 weeks of inpatient psychotherapy. Data will be reported for 7 years of continous study enrollment (2014 - 2021)
  Symptom measure

SECONDARY OUTCOMES:
Relationship Questionnaire 2 (RQ-2) | for each participant: weekly assessment for 8 weeks of inpatient psychotherapy. Data will be reported for 7 years of continous study enrollment (2014 - 2021)
  Attachment measure
Inpatient and day clinic experiences questionnaire (IDES) | for each participant: weekly assessment for 8 weeks of inpatient psychotherapy. Data will be reported for 7 years of continous study enrollment (2014 - 2021)
  measure of self-disclosure and other treatment factors

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Dinger, Prof, Study Chair — University Hospital Heidelberg

IPD SHARING:
Plan to Share IPD: No